CLINICAL TRIAL: NCT05301400
Title: Marginal Bone Loss in Single Implant Restaurations With Three Different Methods
Brief Title: Marginal Bone Loss in Single Implant Restaurations With Different Methods
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Patricia Truchuelo, Clinical Professor and principal investigator, Universidad de León
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ULeon
Record Dates: First submitted 2022-02-26; First posted 2022-03-29 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Overcast implant single restauration (Active Comparator)
  Interventions: Device: Bti Unit
- Cad/cam direct implant restauration (Active Comparator)
  Interventions: Device: Bti Unit
- Cad/cam implant restauration with transepithelial pilar (Active Comparator)
  Interventions: Device: Bti Unit

INTERVENTIONS:
Device: Bti Unit — Comparison with or without the device

SUMMARY:
The investigator is going to measure the marginal bone loss in single implant restaurations with three different methods: direct overcast, milled cad/cam direct to implant restauration and milled cad/cam implant restauration using an transepithelial pilar

DETAILED DESCRIPTION:
The investigator has chosen a statistically significant sample (compared with other similar studies) to analize the bone marginal loss in different types of restauration with single dental implants

ELIGIBILITY:
Inclusion Criteria:

* patients with single implants restaurations treated in Leon University

Exclusion Criteria:

* pregnant
* mayor heath issues
* patients who do not agree to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of marginal loss in single dental implants | 6 months
  To evaluate the vertical loss of bone in milimiters around the implant

SECONDARY OUTCOMES:
Number of Implants with Prosthetic complications | 6 months
  The investigator is going to analyze if there is porcelain chipping (yes or not) and screw loosening (yes or not)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Seco, Study Director — Universidad de León
Locations (1):
- Universidad de Leon, León, Leon, Spain

IPD SHARING:
Plan to Share IPD: Yes
Bone marginal loss
Supporting Information: Study Protocol, SAP, ICF, CSR

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT05301400/Prot_000.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT05301400/ICF_001.pdf